CLINICAL TRIAL: NCT01451957
Title: Fatty Acid Metabolism and Insulin Sensitivity After Exercise in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 03-0165
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: exercise; fatty acid metabolism; insulin sensitivity
MeSH Terms: conditions — Obesity; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): 90 min exercise on Day 1
  Interventions: Other: Exercise - caloric balance
- Sedentary Control (Experimental): Subjects remain sedentary on Day 1 and will either consume a hyper-caloric or a caloric balanced diet
  Interventions: Other: No Exercise - hyper-caloric diet; Other: No exercise - caloric balance

INTERVENTIONS:
Other: Exercise - caloric balance — 90 min exercise on Day 1 with meals afterward resulting in caloric balance for the day (i.e.; extra kcals provided to account for energy expended during exercise)]
  Arms: Exercise
Other: No Exercise - hyper-caloric diet — Subjects remain sedentary on Day 1 and they ingest meals that are identical to those ingested on the day they performed exercise (i.e.; more calories ingested than expended because no exercise performed).
  Arms: Sedentary Control
Other: No exercise - caloric balance — Subjects remain sedentary on Day 1 and they ingest a similar proportion of macronutrients however, the total calories ingested will be lower than the other two trials, resulting in caloric balance for the day.
  Arms: Sedentary Control

SUMMARY:
Alterations in fatty acid mobilization and oxidation may be primary adaptations responsible for the improvements in metabolic health after a single session of endurance exercise. The investigators will determine the effect of a single session of endurance exercise on whole-body fatty acid mobilization and oxidation, IMTG concentration and the expression of factors that regulate these processes in skeletal muscle of 11 women with abdominal obesity (age: 18-45y). In addition, the investigators will evaluate how these factors, and exercise, effect insulin signalling and insulin sensitivity. Every effort will be made to recruit subjects from ethnic and minority groups. Before participating in the study, subjects will be informed of all the procedures and potential risks, and they will sign an informed consent form approved by The University of Michigan Institutional Review Board. Eligible volunteers will participate in three separate trials, in a randomized order. In two trials subjects will eat exactly the same amount of calories, except in one trial they will exercise (eucaloric + exercise) and in the other trial they will remain sedentary (hypercaloric). In a third trial subjects will again remain sedentary but instead they will ingest appropriate calories to maintain caloric balance (eucaloric + sedentary). By doing this the investigators are also able to investigate the effect of acute caloric perturbations on insulin sensitivity, because it is possible that the enhanced insulin sensitivity evident after exercise, as compared to the sedentary state, is due to caloric deficit and not the exercise bout, per se.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal; Body mass index 30-40 kg/m2; Waist circumference >88 cm

Exclusion Criteria:

* Evidence of metabolic or cardiovascular disease; Pregnancy; Hyperlipidemia (fasting plasma triglyceride concentration > 150 mg/dl); Hematocrit < 34%; Undertaking regular exercise (i.e., >2 times/week)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2003-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 3 hours
  frequently sampled intravenous glucose tolerance test(FSIVGTT)will be done to assess insuiln sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Michigan Clincal Research Unit, Ann Arbor, Michigan, United States